CLINICAL TRIAL: NCT00972920
Title: Transversus Abdominis Plane (TAP) Block for Gynaecological Laparotomies - a Comparison of Ultrasound-guided Block and Blind Technique
Brief Title: TAP Block for Gynaecological Laparotomies - a Comparison of Ultrasound-guided Block and Blind Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Health and Social Care Trust (Other Government)
Responsible Party: Principal Investigator, Dr. Pavel Michalek, Locum Consultant Anaesthetist, Northern Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09/NIR03/45
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Laparotomy
Keywords: Transversus abdominis plane; Acute pain service; Ultrasound
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blind TAP block (Active Comparator): TAP block technique as first described by McDonnell. Sterile field obtained with chlorhexidine wash and use of sterile gloves. Identification of triangle of Petit just above iliac crest and between external oblique and latissimus dorsi muscles. Insertion of regional anaesthesia needle perpendicular to skin, and its advancement until sensation of two 'pops' indicating advancement of needle through both external oblique and internal oblique muscle layers.
  After confirmation of negative aspiration the local anaesthetic is injected slowly, (1mg/kg of levobupivacaine), concentration 2.5 mg/mL. Repeat procedure bilaterally (to a maximum dose of 2mg/kg of levobupivacaine).
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- Ultrasound-guided TAP block (Active Comparator): Technique as described by Hebbard. Sterile field obtained with chlorhexidine wash and use of sterile gloves. Ultrasound probe covered with sterile sheath.
  Identification of triangle of Petit with USS probe perpendicular to skin. Insertion of regional anaesthesia needle transversely to the probe, using in-plane (IP) technique, moving posteriorly. Advancement of the needle under ultrasound control until its tip is located between internal oblique and transversus abdominis muscle layers.
  Interventions: Procedure: Transversus abdominis plane (TAP) block

INTERVENTIONS:
Procedure: Transversus abdominis plane (TAP) block — Application of local anaesthetic solution (LA) levo-bupivacaine (dose 1mg/kg for each side, concentration 2.5 mg/mL) between internal oblique abdominis muscle and transversus abdominis muscle on both sides.
  Other Names: TAP block

SUMMARY:
Transversus abdominis plane (TAP) block is an application of local anaesthetic solution into the plane between internal oblique and transversus abdominis muscles at the triangle of Petit located superiorly to the iliac crests bilaterally. Anterior divisions of segmental spinal nerves, which provide innervation to the abdominal wall, run inside this compartment. TAP block been shown to provide good postoperative pain relief following surgical laparotomies, gynaecological laparotomies, appendicectomies, inguinal hernia repairs and open prostatectomies. The goal of this study is to compare the effect of blind and ultrasound-guided TAP block on postoperative pain relief and morphine consumption following to gynaecological laparotomies. Null research hypothesis for the study is that there is no difference between the performance (as defined by morphine consumption and patient satisfaction/ pain scores) of the TAP block procedure via 'blind' or ultrasound guided techniques for gynaecological laparotomies.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block is an application of local anaesthetic solution into the plane between internal oblique and transversus abdominis muscles at the triangle of Petit located superiorly to the iliac crests bilaterally. Anterior divisions of segmental spinal nerves, which provide innervation to the abdominal wall, run inside this compartment. The TAP block has been shown to provide good postoperative pain relief following surgical laparotomies, gynaecological laparotomies, appendicectomies, inguinal hernia repairs and open prostatectomies. It also reduces the post operative morphine consumption seen after such procedures. This allows a more comfortable recovery with reduced incidence of nausea and vomiting, as well as potentially earlier mobilisation and discharge.

Currently the technique employed is that first described by Mc Donnell. This involves a blind 'two pop' technique signifying the needle passing through the two muscle layers. On detection of these two pops the local anaesthetic is injected into this plane between the muscle layers. It is the anaesthetising of the nerves in this muscle plane that aides post operative pain relief for as much as 24 hours. TAP nerve blocks have become common practice due to the very low reported complication rate occurring while using the 'blind technique'. Such complications are minor in themselves. It is our hope that these complications will be further reduced with the use of an ultrasound guided technique. The use of an ultrasound machine would allow the direct visualisation of the needles progress through the tissues and muscle layers. It would confirm the correct position during infiltration of local anaesthetic and prevent inadvertent puncturing of organs or entry to the abdominal space.

Studies have shown that in other commonly used nerve blocks, the introduction of an ultrasound guided technique has improved the efficacy of the nerve block itself. We hope to show a similar trend when using an ultrasound guided technique in the insertion of a TAP block. Trials are underway comparing different dosage and volume regimes, but to our knowledge no other trial is comparing the use of an ultrasound machine to the conventional 'blind' technique in order to assess pain relief and morphine consumption post operatively.

Only recently have ultrasound machines become commonplace in anaesthetic departments, and we feel this research will show their valuable contribution to patient comfort in this subgroup of patients undergoing abdominal gynaecological procedures. We wish to assess whether we can achieve better patient satisfaction, less morphine consumption and ultimately shorter hospital stay with an ultrasound technique compared to a blind technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA status I-III
* Age 18-89 years
* Gynaecological laparotomies with a need for extensive postoperative analgesia.

Exclusion Criteria:

* Patient refusal
* Age less than 18 years or more than 89 years
* ASA status IV or V
* Patients with known reaction to local anaesthetics

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Total consumption of morphine for PCA within the first 12, 24 and 48 hours | 12, 24, 48 hours

SECONDARY OUTCOMES:
Length of High Dependency Unit (recovery) stay | once at discharge
Length of hospital stay | Once at discharge
Visual Analog Scale (VAS) reading | 30min after operation and then at 1hr, 2hrs, 4hrs, 6hrs, 12hrs, 24hrs, 48 hrs
Patient satisfaction | 12, 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Michalek, MD,PhD,DESA, Principal Investigator — Antrim Area Hospital, Northern HSC Trust
Locations (1):
- Antrim Area Hospital, Antrim, Co. Antrim, United Kingdom

REFERENCES:
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039